CLINICAL TRIAL: NCT06105671
Title: Physiological Responses to U-LABA/ICS With Emphasis on Exercise Performance in Well-Trained Individuals, Formoterol
Brief Title: U-LABA/ICS Effects on Exercise Performance, Formoterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morten Hostrup, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FOR
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Exercise Performance
MeSH Terms: interventions — Budesonide, Formoterol Fumarate Drug Combination; Formoterol Fumarate; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Symbicort - usual care (Experimental): Participants are administered Formoterol + Budesonide from an inhaler device testing. In addition, participants are administered a placebo capsule, which is taken orally.
  Interventions: Drug: Symbicort
- Formoterol - inhalation (Experimental): Participants are administered Formoterol from an inhaler device testing. In addition, participants are administered a placebo capsule, which is taken orally.
  Interventions: Drug: Formoterol
- Formoterol - oral (Experimental): Participants are administered a Formoterol capsule, which is taken orally. In addition, participants are administered placebo from an inhaler device.
  Interventions: Drug: Formoterol
- Placebo (Placebo Comparator): Participants are administered placebo from an inhaler device testing and a placebo capsule.
  Interventions: Drug: Placebo
- Mannitol-test (Experimental): Participants are administered Bronchitol from an inhaler device testing.
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Symbicort — Participants are administered 54 μg Formoterol and 1920 μg Budesonide
  Arms: Symbicort - usual care
Drug: Formoterol — Participants are administered 54 μg Formoterol from an inhaler device
  Arms: Formoterol - inhalation
Drug: Formoterol — Participants are administered 120 μg Formoterol in a capsule, which is taken orally
  Arms: Formoterol - oral
Drug: Placebo — Participants are administered placebo
  Arms: Placebo
Drug: Mannitol — Participants are administered 600 mg Bronchitol
  Arms: Mannitol-test

SUMMARY:
The purpose of the project is to investigate exercise performance in well-trained individuals in a crossover design following varying degrees of bronchodilation/constriction intervention using current standard procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Physically active >5 hours a week
* Maximum oxygen uptake classified as high or very high

Exclusion Criteria:

* Diagnosed with severe asthma and been in treatment with long-acting beta2-agonist/corticosteroid
* ECG abnormality
* FEV1/FVC ratio < 0,7 determined with spirometry
* Chronic illness determined to be a potential risk for participant during the study
* In chronic treatments with medication that may interfere with study results
* Pregnancy
* Smoker
* Blood donation during the past 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Power output during time trial | Through study completion, an average on 4 weeks
  Mean power output measured in Watts during a time trial on a bike ergometer

SECONDARY OUTCOMES:
Power output during sprint testing | Through study completion, an average on 4 weeks
  Power output measured in Watts during a sprint on a bike ergometer

OTHER OUTCOMES:
Quadriceps strength | Through study completion, an average on 4 weeks
  Maksimal torque (Nm) achieved during isometric contraction
Forced Expiratory Volume in 1 second (FEV1) | Through study completion, an average on 4 weeks
  FEV1 measured by spirometry
Respiratory muscle function | Through study completion, an average on 4 weeks
  Mouth inspiratory and expiratory pressures against a closed system

CONTACTS AND LOCATIONS:
Overall Officials: Morten Hostrup, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided